CLINICAL TRIAL: NCT04872855
Title: Observational Study to Evaluate the Performance and the Safety of the HLS KneeTec Cementless or Hybrid Fixations in Total Knee Arthroplasty
Brief Title: Observational Study to Evaluate Clinical Performance and Safety in Total Knee Arthroplasty
Status: Terminated | Type: Observational
Why Stopped: the clinical data collected to date are sufficient for regulatory requirements
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP2017-10
Record Dates: First submitted 2021-04-26; First posted 2021-05-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Total Knee Arthroplasty; Knee Disease; Total Knee Replacement; Osteo Arthritis Knee
Keywords: Knee Arthroplasty; Prosthesis; Implants; HLS implants; arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: patient with knee arthroplasty — patient with HLS KneeTec cementless and hybrid fixation prosthesis

SUMMARY:
The aim of this study is to assess the long-term performance and safety of HLS KneeTec cementless and hybrid fixation knee prosthesis when used in standard medical practice.

DETAILED DESCRIPTION:
It is planned to collect prospective and retrospective data from a continuous and exhaustive series of patients in French sites where Total Knee Arthroplasty with HLS Kneetec cementless and hybrid fixation knee prosthesis is performed routinely

All patients treated with HLS KneeTec (cementless or hybrid versions) implant will be included. All eligible patients seen in consultation and who agree to participate in the study should be included, systematically and consecutively, since the initiation of the study.

Patients will be assessed according to the usual practice of the investigator at each participating site before surgery and then at the follow-up (FU) visits as following: 4 months (+/- 2 months); 1 year (+/- 2 months); 5 years (+/- 12 months) and 10 years (+/- 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 - 80 years old at the time of the surgery
* Implanted (or with an indication) with an HLS KneeTec Cementless or hybrid fixation according to the Instructions for Use (IFU)
* Patients agree to consent to collect data from their medical records and agree to answer questionnaires for the purposes of the study.

Exclusion Criteria:

- Patients under guardianship and/or those who, according to the investigator or his delegated research team, will not be able to comply with the study procedures. (e.g. illiteracy, recent psychotic or manic disorders and/or inability to comply with routine follow-up visits.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with HLS KneeTec (cementless or hybrid versions) implant will be included. All eligible patients seen in consultation and who agree to participate in the study should be included, systematically and consecutively, since the initiation of the study
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Evaluation of implant survival in subjects receiving a total knee arthroplasty with the HLS KneeTec cementless and hybrid fixations up to 10 years after the surgery | 10-year
  Kaplan Meier survival rate up to 10 years after the surgery.

SECONDARY OUTCOMES:
Evaluation of clinical performance of the HLS KneeTec cementless and hybrid fixations after the surgery | starting preoperatively up to 10 years
  IKS score
Evaluation of clinical performance of the HLS KneeTec cementless and hybrid fixations after the surgery | 5 and 10 years
  Oxford Knee Score
Radiographic analysis of the HLS KneeTec cementless and hybrid fixations at 4 months, 1, 5 and 10 years minimum | 4 months, 1, 5 and 10 years
  radiological analysis from immediate postoperative up to 10-year FU
Evaluation of safety performance during the surgery up to 10 years after the surgery | starting intraoperatively up to 10-year FU
  Number, severity and casual relationship of procedure or implant-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Franck MABESOONE, MD, Principal Investigator — CH COMPIEGNE
Locations (3):
- France (3):
  - Chu Angers, Angers
  - Clinique Du Parc, Caen
  - Centre Hospitalier Compiegne Noyon, Compiègne